CLINICAL TRIAL: NCT01743768
Title: Clinical Study to Investigate Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of Multiple Doses of the Human GATA-3-specific DNAzyme Solution SB010 in Patients With Mild Allergic Asthma. A Randomised, Double-blind, Parallel, Multicentre, Phase-IIa Study
Brief Title: Safety, Efficacy, PK, and PD Characteristics of Orally Inhaled SB010 in Male Patients With Mild Asthma (Multiple Dose)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sterna Biologicals GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB010/04/2012; 2012-003570-77 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: Antisense oligonucleotide; Asthma; Healthy subjects; Phase 1; Transcription factor GATA-3; Oral inhalation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB010 (Experimental): The drug will be administered in phosphate-buffered saline solution, inhaled over 5 - 10 min, using inhalation device.
  Administered dose: 10 mg hgd40 in 2 mL solution (5.0 mg/mL).
  Initial dose on Day 1 (single-dose PK profile); once daily dose for 28 consecutive days (Days 1 to 28); last inhalation on Day 28 (steady state PK profile).
  Interventions: Drug: SB010
- Placebo (Placebo Comparator): The placebo (phosphate-buffered saline) is administered as a solution, inhaled over 5 - 10 min, using inhalation device.
  Initial dose on Day 1 (single-dose PK profile); once daily dose for 28 consecutive days (Days 1 to 28); last inhalation on Day 28 (steady state PK profile).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB010 — Treatment group (n=19), receiving the active drug substance.
  Other Names: Active drug substance is hgd40
  Arms: SB010
Drug: Placebo — Treatment group (n=19), receiving placebo.
  Other Names: Phosphate-buffered saline
  Arms: Placebo

SUMMARY:
Asthma is a chronic inflammatory bronchial disorder with three distinct components: airway hyper-responsiveness (respiratory hypersensitivity), airway inflammation, and intermittent airway obstruction. One of the characteristics of the disease is an inflammatory reaction of the immune system caused by cytokine production. A substantial number of asthma patients do not satisfactorily respond to steroid therapy and consequently have an unmet medical need for novel targeted therapies with improved specificity, tolerability, and compliance.

Novel therapeutic strategies for the treatment of chronic inflammatory diseases by targeting early disease-causing mechanisms are a promising approach for the treatment of asthma. The transcription factor GATA-3 plays a key role in mediating the asthmatic immune response and has been shown to be necessary and sufficient for the production of cytokines interleukin (IL)-4, IL-5, and IL-13. The active drug substance of the investigational medicinal product SB010 is hgd40. SB010 belongs to a new class of antisense oligonucleotide therapeutics, the 10-23 DNA (deoxyribonucleic acid)zymes (antisense oligonucleotide).

DNAzymes are catalytically active nucleic acids that cleave complementary RNA (ribonucleic acid) molecules. By cleaving GATA-3 mRNA, hgd40 reduces specific cytokine production and thereby reduces key features of allergic airway inflammation. DNAzymes are generated completely by chemical synthesis and can be produced under Good Manufacturing Practice (GMP) controlled conditions. The DNAzymes are not biological drugs, i.e. they are not generated by use of any living organism including cell culture or bacteria. The molecules are highly water-soluble and will be applied as solution directly in their synthesized form.

This proof-of-concept study will evaluate the safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of inhaled SB010 in male patients with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male Caucasian patients aged ≥ 18 and ≤ 60 years.
2. Clinical diagnosis of mild asthma (according to GINA guidelines 2008 update) for at least 6 months prior to screening. No concomitant asthma treatment. except inhaled short-acting bronchodilators.
3. Screening FEV1 value of FEV1 ≥ 70 % of the predicted normal value (ECSC) after a wash out of at least 6 hours for inhaled short-acting bronchodilators,
4. Patient must demonstrate sufficient induced sputum production.
5. Positive skin prick test (skin reactivity) to common aeroallergens (e.g. animal epithelia, dust mite).
6. Patient must demonstrate positive allergen-induced early- and late-phase airway bronchoconstriction.
7. At all timepoints before AC and MCh, patients must show FEV1 not below 65 % predicted.
8. Presence of sputum eosinophils either before or after screening allergen challenge (first or second induced sputum).
9. Patient has been informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which he may be exposed, and has given written consent to participation in the trial prior to trial start and any trial-related procedure.
10. Patient is able to understand and give written informed consent and has signed a written informed consent form approved by the Investigator's Research Ethics Board.
11. Non-smokers or ex-smokers who had stopped smoking for at least 1 year prior to start of the clinical study with < 10 pack years.
12. Ability to inhale in an appropriate manner (patients will be trained to inhale from the AKITA2 APIXNEB® device with a placebo medication at the screening visit).
13. Only men who do not want to father children for six months after the last dose of SB010 will be included into this study.

Exclusion Criteria:

1. Presence of clinically significant diseases other than asthma (cardiovascular, renal, hepatic, gastrointestinal, haematological, neurological, genitourinary, autoimmune, endocrine, metabolic, etc.), which, in the opinion of the investigator, may either put the patient at risk because of participation in the trial, or diseases which may influence the results of the study or the patient's ability to take part in it.
2. Presence of relevant pulmonary diseases or history of thoracic surgery, such as:

   * known active tuberculosis,
   * History of interstitial lung or pulmonary thromboembolic disease,
   * Pulmonary resection during the past 12 months,
   * History of status asthmaticus,
   * History of bronchiectasis secondary to respiratory diseases (e.g. cystic fibrosis, Kartagener's syndrome, etc.),
   * History of chronic bronchitis, emphysema, allergic bronchopulmonary aspergillosis or respiratory infection within the 4 preceding weeks of the first morning IMP administration.
3. Patients on concomitant treatments, except for inhaled short-acting bronchodilators as judged by the investigator.
4. Use of short-acting ß2-agonists 6 hours before study visits 2, 3, 4, 5, 11, and 12.
5. Hospitalisation or emergency room treatment for acute asthma in the 6 months prior to screening, between screening and the start of the treatment period.
6. Intubation (ever) or hospitalisation for longer than 24 hours for the management of an asthma exacerbation within the preceding 6 months of the screening visit.
7. History or current evidence of clinically relevant allergies or idiosyncrasy to drugs.
8. History of allergic reactions to any active or inactive ingredients of the nebuliser solution.
9. ECG abnormalities of clinical relevance.
10. Subjects with a resting heart rate < 45 bpm, systolic blood pressure < 100 mmHg, diastolic blood pressure < 60 mmHg.
11. Proneness to orthostatic dysregulation, fainting, or blackouts.
12. History of malignancy within the past 5 years, except excised basaliomas.
13. Clinically relevant abnormalities in clinical chemical, haematological or in any other laboratory variables as judged by the investigator.
14. Clinically relevant acute infections in the last 4 weeks preceding AC.
15. Clinically relevant chronic infections.
16. Positive results in any of the virology tests of acute or chronic infectious human immunodeficiency virus (HIV) and hepatitis B/C virus infections.
17. Positive drug screen.
18. Abuse of alcohol or drugs.
19. Positive cotinine test.
20. Treatment with any known enzyme inducing or inhibiting agents (St. John's Wort (Johanniskraut), barbiturates, phenothiazines, cimetidine, ketoconazole etc.) within 30 days before first administration of trial medication or during treatment period of the trial.
21. Use of any prohibited concomitant medication within 2 weeks (for biologics: 6 months or 10 times the elimination half-life of the respective drug) before first trial medication administration or within < 10 times the elimination half-life of the respective drug, or the duration of the pharmacodynamic effect, whatever is longer, or anticipated concomitant medication during the treatment period.
22. Consumption of any enzyme inducing or inhibiting aliments and beverages (e.g. broccoli, Brussels sprout, grapefruit, grapefruit juice, star fruit etc.) within 14 days prior to the first trial medication administration and during the treatment period of the trial.
23. Consumption of any caffeine-containing product 6 hours before first procedure at each study visit.
24. Surgery of the gastrointestinal tract which may interfere with drug absorption of swallowed fraction (Note: this is not applicable for minor abdominal surgery such as appendectomy or herniotomy).
25. Blood donation within the last 30 days before screening.
26. Planned donation of germ cells, blood, organs or bone marrow during the course of the trial or within 6 months thereafter.
27. Participation in another clinical trial with an investigational drug or device within the last month or within 10 times the half-life of the respective drug. For biologics the minimum period is at least 6 months or the time of duration of the pharmacodynamic effect or 10 times the half-life of the respective drug before inclusion in this trial.
28. Lack of ability or willingness to give informed consent or inability to cooperate adequately.
29. Anticipated non-availability for trial visits/procedures.
30. Vulnerable subjects (e.g., persons kept in detention).
31. Employee at the investigational site, relative or spouse of the investigator.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in late phase response after allergen challenge (AC), following multiple doses of inhaled SB010 | Day -1 and Day 28 (monitoring for 7 h after AC).
  After 28 days of treatment with SB010 or placebo, patients will undergo allergen bronchoprovocation [allergen challenge (AC)]. The results from AC on Day 28 will be compared to results obtained on Enrolment (Day -1).
  Allergen for AC will be selected based on skin prick test performed at Screening. The dose of selected allergen will be determined based on skin prick dilution test.
  After the AC, serial spirometry will be used to assess the influence of inhaled SB010 on the area under the Forced Expiratory Volume in 1 second (FEV1) curve during the late asthma response (LAR, 4 - 7 hours); measurement time points will be at 4, 5, 6, and 7 hours after AC.
  The spirometric parameters FEV1 and forced vital capacity (FVC), obtained during pulmonary function testing, will be used to derive the primary efficacy variable AUC4-7 FEV1.

SECONDARY OUTCOMES:
Number of patients with adverse events after multiple doses of inhaled SB010 | Screening examination (Day -56 to -14 before first drug administration); Study period (Day 1 to 28); Follow-up visit (Day 88±4); Maximum of 149 days for a particular subject.
  Investigate occurrence of adverse events.
Number of patients with changes in vital signs after multiple doses of inhaled SB010 | Screening examination (Day -56 to -14 before first drug administration); Study period (Day 1 to 28); Follow-up visit (Day 88±4); Maximum of 149 days for a particular subject.
  Investigate any change in vital signs.
Number of patients with changes in electrocardiogram (ECG) after multiple doses of inhaled SB010 | Screening examination (Day -56 to -14 before first drug administration); Study period (Day 1 to 28); Follow-up visit (Day 88±4); Maximum of 149 days for a particular subject.
  Investigate any change in electrocardiogram (ECG).
Number of patients with changes in safety laboratory tests after multiple doses of inhaled SB010 | Screening examination (Day -56 to -14 before first drug administration); Study period (Day 1 to 28); Follow-up visit (Day 88±4); Maximum of 149 days for a particular subject.
  Investigate any change in safety laboratory tests (clinical chemistry, coagulation, immune monitoring, hematology, urine analysis).
Number of patients with changes in spirometry laboratory tests (FEV1, FVC) after multiple doses of inhaled SB010 | Screening examination (Day -56 to -14 before first drug administration); Study period (Day 1 to 28); Follow-up visit (Day 88±4); Maximum of 149 days for a particular subject.
  Investigate the number of patients with changes in spirometry laboratory tests [Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC)], after multiple doses of inhaled SB010.

OTHER OUTCOMES:
Area under the FEV1 curve during early phase response (0 - 3 hours) after allergen challenge (AC) | Screening (Day -54 to -15); Enrolment (Day -1); Study period (Day 28).
  Serial spirometry will be performed to assess the influence of multiple doses of inhaled SB010 on the area under the FEV1 curve in the early phase response (EAR, 0-3 hours) following allergen challenge (AC). The measurement time points are 10, 20, 40, 60, 120, and 180 min after AC.
Allergen-induced airway responsiveness (PC20 methacholine) | Screening (Day -56 to -17); Baseline (Day 0); Endpoint assessment (Day 29).
  Investigate the influence of multiple doses of inhaled SB010 on allergen-induced airway responsiveness. PC20# will be assessed in subgroups.
  #PC20=Provocative concentration of a substance ( methacholine) causing a 20% fall in FEV1.
Fractionated exhaled nitric oxide (FeNO) | Enrolment (Day -1); Baseline (Day 0); Study period (Day 1, 13±1, 28); Endpoint assessment (Day 29); Follow-up assessment (Day 88±4).
  Investigate the impact of multiple doses of inhaled SB010 on levels of fractionated exhaled nitric oxide (FeNO) .
Systemic biomarkers | Enrolment (Day -1); Baseline (Day 0); Study period (Day 28); Endpoint assessment (Day 29).
  Investigate the influence of multiple doses of inhaled SB010 on systemic biomarkers in plasma, including IL-4, IL-5, IL-10, IL-13, IFN-gamma, Periostin.
Sputum parameters | Screening (Day -56 to -17; Day -53 to -14); Baseline (Day 0); Study period (Day 26±1); Endpoint assessment (Day 29).
  Investigate the influence of multiple doses of inhaled SB010 on sputum parameters (differential cell counts, soluble mediators including tryptase, ECP and Th1/Th2 cytokines as well as explorative mRNA analysis), and sputum eosinophils.
Area under the plasma concentration versus time curve (AUC0-infinity) of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.
Dose-normalized area under the plasma concentration versus time (AUC0-infinity) of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.
Concentration maximum (Cmax) of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.
Dose-normalized concentration maximum (Cmax) of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.
Time of maximum concentration (tmax) of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.
Apparent terminal elimination half-life of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.
Area under the concentration-time curve until the last sampling time (tlast) with a quantifiable concentration (AUC0-tlast) of SB010 | Study period (Day 1 and Day 28).
  The pharmacokinetic parameter will be calculated from plasma concentrations of hgd40 using non-compartmental procedures after a single dose on Day 1 and after repeated dosing at steady state on Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, Prof MD, Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine, Hannover, Germany
Locations (7):
- Germany (7):
  - Charité Research Organisation GmbH, Berlin
  - Clinical Research Centre RespiratoryMedicine (IKF), Frankfurt
  - Inamed GmbH, Gauting
  - Pulmonary Research Institute (PRI), Großhansdorf
  - Clinical Airway Research Fraunhofer Institute for Toxicology and Experimental Medicine (ITEM), Hanover
  - Johannes Gutenberg University Medical Clinic III for Hematology, Oncology and Pneumology, Mainz
  - insaf - Respiratory Research Institute GmbH, Wiesbaden

REFERENCES:
- [Derived] Krug N, Hohlfeld JM, Kirsten AM, Kornmann O, Beeh KM, Kappeler D, Korn S, Ignatenko S, Timmer W, Rogon C, Zeitvogel J, Zhang N, Bille J, Homburg U, Turowska A, Bachert C, Werfel T, Buhl R, Renz J, Garn H, Renz H. Allergen-induced asthmatic responses modified by a GATA3-specific DNAzyme. N Engl J Med. 2015 May 21;372(21):1987-95. doi: 10.1056/NEJMoa1411776. Epub 2015 May 17. PMID 25981191